CLINICAL TRIAL: NCT06709794
Title: Evaluating the Effect of Automatic Plan Assignment and Enhanced Outreach of Marketplace Take-up
Acronym: MAPS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Covered California (Other Government)
Responsible Party: Principal Investigator, Emory Wolf, Assistant Deputy Director, Evaluation & Research, Covered California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CCA-MAPS-2024
Record Dates: First submitted 2024-11-18; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Outreach Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): A control group that receives a standard eligibility notice informing them of their eligibility for marketplace coverage.
- Enhanced Outreach (Experimental): A treatment group that receives a standard eligibility notice informing them of their eligibility for marketplace coverage and an informational flyer describing what Covered California is, the availability of financial assistance, and information on benefit design and private insurance terminology, such as deductibles and copays.
  Interventions: Behavioral: Informational flyer
- Pre-Selected Plan (Experimental): A treatment group that receives a modified eligibility notice that includes information on the pre-selected lowest-cost silver health insurance plan with a personalized quote for their net premium amount, as well as the informational flyer.
  Interventions: Behavioral: Modified eligibility notice with plan information

INTERVENTIONS:
Behavioral: Informational flyer — In addition to a standard eligibility notice informing participants of their eligibility for marketplace coverage, they receive an informational flyer describing what Covered California is, the availability of financial assistance, and information on benefit design and private insurance terminology, such as deductibles and copays
  Arms: Enhanced Outreach
Behavioral: Modified eligibility notice with plan information — a modified eligibility notice that includes information on the pre-selected lowest-cost silver health insurance plan with a personalized quote for their net premium amount in addition to the informational flyer and instead of a standard eligibility notice
  Arms: Pre-Selected Plan

SUMMARY:
Facilitated enrollment offers a potential solution to some administrative burdens and choice frictions that may produce incomplete take-up of marketplace coverage. Because Covered California, California's ACA individual marketplace, and Medi-Cal, California's Medicaid program, share an eligibility system, Covered California has the ability to identify individuals who are eligible for marketplace coverage upon losing Medicaid eligibility.

This evaluation will compare the effectiveness of facilitated enrollment strategies, including personalized plan pre-selection and personalized quotes of net premiums, to other enhanced, but general outreach tactics, on marketplace take-up among individuals losing Medi-Cal coverage.

ELIGIBILITY:
Inclusion Criteria:

* Individual in a single-member household
* Discontinued from Medi-Cal
* Eligible for Covered California program
* Ineligible for APTCs on initial application
* Did not attest to planning to file taxes within their Covered California application

Exclusion Criteria:

* Consumer case is no longer active within the application system
* Consumer is already actively enrolled in a marketplace plan
* Consumer has already restored Medi-Cal eligibility
* A consumer's Special Enrollment Period has ended
* Consumer is no longer listed as a single-member household
* Consumer was procedurally denied from Medi-Cal coverage due to no response
* Consumers has a MAGI Medi-Cal income less than 138% of the Federal Poverty Level (FPL)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment | within calendar year since the loss of Medicaid
  a binary indicator for whether a consumer has at least one month of effectuated coverage a Covered California plan that started within the 90 days of their Special Enrollment Period (SEP) following loss of Medi-Cal coverage

SECONDARY OUTCOMES:
Tenure | within 1-2 years after treatment assignment
  Tenure with Covered California (measured in months)
Uninsured | within 1-2 years from the treatment assignment
  A binary indicator for whether someone self-reported being uninsured while filing their taxes;
Consumer engagement | within 90 days from the treatment assignment
  A binary indicator for consumer engagement including calls to service center, creation of and logins to user account, plan shopping on the website, agent delegation after eligibility determination;
Office visit | during 1-2 years since the treatment assignment
  A binary indicator for whether someone had an office visit to the medical practitioner during 1-2 years since the intervention;
Prescription filled | during 1-2 years since the treatment assignment
  A binary indicator for whether someone had a prescription drug fill during 1-2 years since the intervention;
Emergency room visit | during 1-2 years since the treatment assignment
  A binary indicator for whether someone had an emergency room or department visit during 1-2 years since the intervention
Hospital admission | 1-2 years before and during 1-2 years after the treatment assignment
  A binary indicator for whether someone had a hospital admission 1-2 years before and during 1-2 years since the intervention
Out-of-pocket health care spending | during 1-2 years since the treatment assignment
  Total out-of-pocket spending for the 1-2 years since the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Covered California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT06709794/Prot_SAP_000.pdf